CLINICAL TRIAL: NCT03584048
Title: Charlotte Retention in Care Study - Clinical Decision Support System Prompts
Brief Title: Charlotte Retention in Care Study
Status: Completed | Type: Observational
Sponsor: Epividian (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: HO-18-19095
Record Dates: First submitted 2018-05-17; First posted 2018-07-12 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2019-10

CONDITIONS: HIV I Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 17 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-1: HIV-1+, males, females, transgender, ≥18 years of age, residing in the Charlotte Metropolitan Area and with at least a single entry in the EHR in the last 2 years.
  Interventions: Other: Alert to provider

INTERVENTIONS:
Other: Alert to provider — Providers receive alerts of sub-optimal patient attendance using 4 rules.

SUMMARY:
The objective of the Charlotte Retention in Care study is to assess if clinical decision support systems (CDSS) that produce standardized alerts for measures of retention in care across clinics in the city of Charlotte, North Carolina have the ability to increase retention in care measures within clinics and in surveillance reports.

DETAILED DESCRIPTION:
Multiple Charlotte HIV Clinic providers are participating. "Primary" HIV provider will be defined as the primary physician or advanced care practitioner following a patient, as recorded in their respective Electronic Health Record (EHR) system and identified through CHORUS, a Clinical Decision Support System (CDSS) developed by Epividian. The CDSS will track patient case status as active or inactive (loss to follow-up, transferred medical care, or deceased). Providers will be informed of the study and sites will be contracted to participate in this collaborative research study. This study was approved by the Advarra Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1+
* Any gender
* 18 years old or older
* Residing in the Charlotte, North Carolina metropolitan area
* At least a single entry in the EHR in the last 2 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIV-1+, males, females, transgender, ≥18 years of age, residing in the Charlotte Metropolitan Area and with at least a single entry in the EHR in the last 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Engagement level | 12 months, 01-Nov-2018 to 31-Oct-2019
  Pre and post-baseline engagement level. Engagement level is defined as patients with 0, 1, or 2+ visits to physician (identified as a visit that included the collection of 1 viral load and/or 1 CD4 count lab test).

SECONDARY OUTCOMES:
Kept appointment | 12 months, 01-Nov-2018 to 31-Oct-2019
  Pre and post-baseline "kept appointment rate", the proportion of patients who attended their scheduled office visits.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leonard, MD, Principal Investigator — Atrium Health (Carolinas HealthCare System)
Locations (4):
- United States (4):
  - Atrium Health, Charlotte, North Carolina
  - Amity Group Foundation, Charlotte, North Carolina
  - Ballantyne Family Medicine, Charlotte, North Carolina
  - Rosedale Medical, Huntersville, North Carolina

IPD SHARING:
Plan to Share IPD: No
No Protected Health Information (PHI) is shared outside of clinic. De-identified data available only to authorized researchers via Epividian Clinical Advisory Board approval.

REFERENCES:
- [Background] Bakken S. An informatics infrastructure is essential for evidence-based practice. J Am Med Inform Assoc. 2001 May-Jun;8(3):199-201. doi: 10.1136/jamia.2001.0080199. PMID 11320064
- [Background] Bates DW, Gawande AA. Improving safety with information technology. N Engl J Med. 2003 Jun 19;348(25):2526-34. doi: 10.1056/NEJMsa020847. No abstract available. PMID 12815139
- [Background] Bakken S, Cimino JJ, Hripcsak G. Promoting patient safety and enabling evidence-based practice through informatics. Med Care. 2004 Feb;42(2 Suppl):II49-56. doi: 10.1097/01.mlr.0000109125.00113.f4. PMID 14734942
- [Background] Jenders RA, Osheroff JA, Sittig DF, Pifer EA, Teich JM. Recommendations for clinical decision support deployment: synthesis of a roundtable of medical directors of information systems. AMIA Annu Symp Proc. 2007 Oct 11;2007:359-63. PMID 18693858
- [Background] Schulman J, Kuperman GJ, Kharbanda A, Kaushal R. Discovering how to think about a hospital patient information system by struggling to evaluate it: a committee's journal. J Am Med Inform Assoc. 2007 Sep-Oct;14(5):537-41. doi: 10.1197/jamia.M2436. Epub 2007 Jun 28. PMID 17600095
- [Background] Patel V, Abramson EL, Edwards A, Malhotra S, Kaushal R. Physicians' potential use and preferences related to health information exchange. Int J Med Inform. 2011 Mar;80(3):171-80. doi: 10.1016/j.ijmedinf.2010.11.008. Epub 2010 Dec 14. PMID 21156351
- [Background] Middleton B, Hammond WE, Brennan PF, Cooper GF. Accelerating U.S. EHR adoption: how to get there from here. recommendations based on the 2004 ACMI retreat. J Am Med Inform Assoc. 2005 Jan-Feb;12(1):13-9. doi: 10.1197/jamia.M1669. Epub 2004 Oct 18. PMID 15492028
- [Background] Garg AX, Adhikari NK, McDonald H, Rosas-Arellano MP, Devereaux PJ, Beyene J, Sam J, Haynes RB. Effects of computerized clinical decision support systems on practitioner performance and patient outcomes: a systematic review. JAMA. 2005 Mar 9;293(10):1223-38. doi: 10.1001/jama.293.10.1223. PMID 15755945
- [Background] Poon EG, Wald J, Bates DW, Middleton B, Kuperman GJ, Gandhi TK. Supporting patient care beyond the clinical encounter: three informatics innovations from partners health care. AMIA Annu Symp Proc. 2003;2003:1072. PMID 14728575
- [Background] Bakken S, Roberts WD, Chen E, Dilone J, Lee NJ, Mendonca E, Markatou M. PDA-based informatics strategies for tobacco use screening and smoking cessation management: a case study. Stud Health Technol Inform. 2007;129(Pt 2):1447-51. PMID 17911954
- [Background] Bindoff IK, Tenni PC, Peterson GM, Kang BH, Jackson SL. Development of an intelligent decision support system for medication review. J Clin Pharm Ther. 2007 Feb;32(1):81-8. doi: 10.1111/j.1365-2710.2007.00801.x. PMID 17286791
- [Background] Dickey J, Girard DE, Geheb MA, Cassel CK. Using systems-based practice to integrate education and clinical services. Med Teach. 2004 Aug;26(5):428-34. doi: 10.1080/01421590410001730967. PMID 15369883
- [Background] Grant RW, Wald JS, Poon EG, Schnipper JL, Gandhi TK, Volk LA, Middleton B. Design and implementation of a web-based patient portal linked to an ambulatory care electronic health record: patient gateway for diabetes collaborative care. Diabetes Technol Ther. 2006 Oct;8(5):576-86. doi: 10.1089/dia.2006.8.576. PMID 17037972
- [Background] Hsieh TC, Kuperman GJ, Jaggi T, Hojnowski-Diaz P, Fiskio J, Williams DH, Bates DW, Gandhi TK. Characteristics and consequences of drug allergy alert overrides in a computerized physician order entry system. J Am Med Inform Assoc. 2004 Nov-Dec;11(6):482-91. doi: 10.1197/jamia.M1556. Epub 2004 Aug 6. PMID 15298998
- [Background] Lester WT, Ashburner JM, Grant RW, Chueh HC, Barry MJ, Atlas SJ. Mammography FastTrack: an intervention to facilitate reminders for breast cancer screening across a heterogeneous multi-clinic primary care network. J Am Med Inform Assoc. 2009 Mar-Apr;16(2):187-95. doi: 10.1197/jamia.M2813. Epub 2008 Dec 11. PMID 19074304
- [Background] Lester WT, Grant R, Barnett GO, Chueh H. Facilitated lipid management using interactive e-mail: preliminary results of a randomized controlled trial. Stud Health Technol Inform. 2004;107(Pt 1):232-6. PMID 15360809
- [Background] Lester WT, Grant RW, Barnett GO, Chueh HC. Randomized controlled trial of an informatics-based intervention to increase statin prescription for secondary prevention of coronary disease. J Gen Intern Med. 2006 Jan;21(1):22-9. doi: 10.1111/j.1525-1497.2005.00268.x. PMID 16423119
- [Background] Cowen M, Halasyamani LK, McMurtrie D, Hoffman D, Polley T, Alexander JA. Organizational structure for addressing the attributes of the ideal healthcare delivery system. J Healthc Manag. 2008 Nov-Dec;53(6):407-18; discussion 419. PMID 19070335
- [Background] Crosson FJ. The delivery system matters. Health Aff (Millwood). 2005 Nov-Dec;24(6):1543-8. doi: 10.1377/hlthaff.24.6.1543. PMID 16284026
- [Background] Doebbeling BN, Chou AF, Tierney WM. Priorities and strategies for the implementation of integrated informatics and communications technology to improve evidence-based practice. J Gen Intern Med. 2006 Feb;21 Suppl 2(Suppl 2):S50-7. doi: 10.1111/j.1525-1497.2006.00363.x. PMID 16637961
- [Background] McGowan JJ, Cusack CM, Poon EG. Formative evaluation: a critical component in EHR implementation. J Am Med Inform Assoc. 2008 May-Jun;15(3):297-301. doi: 10.1197/jamia.M2584. Epub 2008 Feb 28. PMID 18308984
- [Background] Rind DM, Safran C, Phillips RS, Wang Q, Calkins DR, Delbanco TL, Bleich HL, Slack WV. Effect of computer-based alerts on the treatment and outcomes of hospitalized patients. Arch Intern Med. 1994 Jul 11;154(13):1511-7. PMID 8018007
- [Background] Ruland CM, Bakken S. Developing, implementing, and evaluating decision support systems for shared decision making in patient care: a conceptual model and case illustration. J Biomed Inform. 2002 Oct-Dec;35(5-6):313-21. doi: 10.1016/s1532-0464(03)00037-6. PMID 12968780